CLINICAL TRIAL: NCT00417352
Title: Kinematic and Kinetic Profile of Common Tasks for the Development of Design Parameters of an Upper Limb Prosthesis
Brief Title: Study of Compensatory Motion While Using an Upper Limb Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Responsible Party: Stephanie L. Carey, University of South Florida Mechanical Engineering Dept.
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: Compensatory motion
Record Dates: First submitted 2006-12-28; First posted 2007-01-01 (Estimated); Last update posted 2010-08-06 (Estimated); Status verified 2006-12

CONDITIONS: Prosthesis
Keywords: no intervention; bracing restricted forearm and wrist movement; bracing with added mass near elbow; bracing with added mass near wrist
MeSH Terms: interventions — Braces

INTERVENTIONS:
Device: Brace
Device: Added mass

SUMMARY:
Current improvements of the design of the upper limb prosthesis include advanced technology in control systems and electronic circuitry that mimic human motion and improve function of the prosthesis. Often times these improvements require large amounts of power, circuitry and excess mass distally along the prosthesis that may require greater effort from the user. Poor function of an upper limb prosthesis may cause awkward compensatory motion. Aberrant movements, such as these compensatory movements are known to cause greater stress to remaining joints. Amputees are forced to decide if the extra function provided by the advanced electronics is worth carrying the extra mass which may cause fatigue, socket issues and greater stress on the remaining joints. An example is the wrist rotator component of an upper limb prosthesis which may allow greater function and reduce compensatory motion, but adds mass distally, potentially causing greater torques on remaining joints.

GOALS OF THE STUDY:

There are two main goals of this study:

1. to determine the impact of an upper limb prosthesis without a wrist rotator on the compensatory motion and torques in the remaining joints during common tasks
2. to determine the impact of the location (distally or proximally) of a wrist rotator on a upper limb prosthesis on the compensatory motion during common tasks

HYPOTHESES:

1. There will be a statistically significant difference in range of motion of the upper limb joints between healthy subjects, braced subjects and upper limb amputees during four common tasks.
2. There will be a statistically significant difference in joint upper limb joint torques between healthy subjects, braced subjects and upper limb amputees during three common tasks.
3. There will be a statistically significant difference in upper limb angles and joint torques between mass added distally and mass added proximally during common tasks.

DETAILED DESCRIPTION:
PROBLEM STATEMENT:

Current improvements of the design of the upper limb prosthesis include advanced technology in control systems and electronic circuitry that mimic human motion and improve function of the prosthesis. Often times these improvements require large amounts of power, circuitry and excess mass distally along the prosthesis that may require greater effort from the user. Poor function of an upper limb prosthesis may cause awkward compensatory motion. Aberrant movements, such as these compensatory movements are known to cause greater stress to remaining joints. Amputees are forced to decide if the extra function provided by the advanced electronics is worth carrying the extra mass which may cause fatigue, socket issues and greater stress on the remaining joints. An example is the wrist rotator component of an upper limb prosthesis which may allow greater function and reduce compensatory motion, but adds mass distally, potentially causing greater torques on remaining joints.

SYNOPSIS OF CURRENT LITERATURE:

Restricted motion and excess weight of an upper limb prosthesis have been documented as complaints among amputees [1], [2], [3], [4], [5], [6]. Through surveys Atkins et al. determined that amputees would like the wrist component of the prosthesis to perform more movements. This study also listed drinking from a glass and opening a door, top priorities among amputees [7]. This suggests that the wrist component on a prosthetic arm is important.

There are many examples throughout scientific literature showing how kinetic, kinematic and metabolic analyses of gait have lead to the improvement of lower limb prosthetic design criteria [8],[9]. In 2003, Twiste et al. conducted a literature review on rotation and translation of the anatomic joints during prosthetic gait. The abstract from this review mentions that more accurate kinematic gait analysis showing optimized gait patterns could help manufacturers design prosthetic components to mimic these patterns [9]. The effects of mass perturbations on lower limb amputees have been investigated to determine how inertial properties of a prosthesis should be evaluated [10].

There have also been studies involving upper limb motion, but the amount is limited. The range of motion of the upper limb of healthy and braced subjects performing activities of daily living have been recorded and analyzed [11],[12],[13]. These studies have looked at the effect of wrist position, but not on the mass of a wrist component.

GOALS OF THE STUDY:

There are two main goals of this study:

1. to determine the impact of an upper limb prosthesis without a wrist rotator on the compensatory motion and torques in the remaining joints during common tasks
2. to determine the impact of the location (distally or proximally) of a wrist rotator on a upper limb prosthesis on the compensatory motion during common tasks

HYPOTHESES:

1. There will be a statistically significant difference in range of motion of the upper limb joints between healthy subjects, braced subjects and upper limb amputees during four common tasks.
2. There will be a statistically significant difference in joint upper limb joint torques between healthy subjects, braced subjects and upper limb amputees during three common tasks.
3. There will be a statistically significant difference in upper limb angles and joint torques between mass added distally and mass added proximally during common tasks.

METHODS Participants Ten healthy adult volunteers with no history of upper limb injury will participate in this study. Five men and five women will participate. These ten subjects will make up the control group and then will be braced to simulate a below elbow prosthesis. Seven unilateral upper limb amputees will participate.

Testing Protocol An 8 camera infrared Vicon motion analysis system will be used for the collection and analysis of movement data. Nineteen spherical reflective markers will be placed on the boney landmarks of the upper limbs and torso of the subjects to describe segments or local coordinate systems.

A static trial will be collected for each subject to help determine the joint centers. Subject parameters such as body mass, height, and shoulder depth, wrist and hand thickness will be collected for use in calculations. Kinematic data will be collected at 120 Hz.

Subjects will be asked to complete four tasks:

* Drinking from a cup
* Opening a door
* Lifting a 5 lb. box
* Turning a steering wheel ( kinetic analysis of this task will be excluded)

The healthy subjects will complete each task during following interventions: (1) no intervention (2) braced restricting forearm and wrist motion, (3) braced with 96 g (mass of average prosthetic wrist rotator) added near the elbow, (4) braced with 96 g added near the wrist. The amputees will complete interventions (3) and (4) mentioned above without a wrist rotator but simulating the mass of one. Three trials will be collected for each experimental test condition and these trials will be averaged as a representative for each subject. The order of the tests will be randomly assigned for each subject.

Design of Experiment:

This study will look at the effects of the absence of wrist and forearm motion on shoulder, elbow and torso motion during four activities. This study will combine between-subject and within-subject analysis.

Independent factor (between subjects): restriction of wrist and forearm movement (simulating no wrist rotator component on prosthesis)

Levels:

* Control group
* Braced group - simulating a below elbow upper limb prosthesis
* Prosthesis wearing group

Repeated factor (with-in subjects): added mass (simulating the mass of wrist rotator)

Levels:

* No added mass of a wrist rotator
* Mass of a wrist rotator added proximally (near elbow)
* Mass of a wrist rotator added distally (near wrist)

A two-way analysis of variance with one repeated measure will be used to analyze the main effects and the interaction effects.

Data Processing

Shoulder, elbow and torso motions and torques will be computed using a program written in Vicon Bodybuilder language. The positions of the markers placed on the subject will be digitized and torso, upper arm, lower arm and hand segments will be determined. Euler angles will be computed. Inverse dynamics and anthropometrics will be used to compute forces and torques. The following outcome measures will be compared:

* Shoulder abduction and flexion
* Elbow flexion
* Torso bending (L/R)
* Shoulder joint force and torque
* Elbow joint force and torque

The maximum, minimum and range of these outcome measures will be compared between subjects and with-in subjects.

PREDICTED RESULTS/DISCUSSION

Drinking from a cup:

* Braced and prosthesis wearing groups will have greater shoulder abduction to compensate for the lack of forearm rotation and wrist extension.
* Adding the mass (wrist rotator) distally will cause a greater force and torque at the elbow. This increase of forces at the elbow will be greatest in the amputee group due to possible injury to the brachialis at its insertion on the tuberosity of the ulna.

Opening a door:

* Braced and prosthesis wearing groups will have greater shoulder abduction to compensate for the lack of forearm rotation and wrist extension. These groups may also compensate by the bending the trunk instead of increasing shoulder abduction.
* Due to the increased shoulder range of motion in the coronal plane, the braced and prosthesis wearing group will have a greater torque at the shoulder joint. This increase of shoulder joint torque will increase when the mass (wrist rotator) is added distally due to the increase in the lever arm.

Lifting a 5 lb. box:

* This task will require minimal wrist deviation, wrist flexion/extension and minimal forearm rotation. It is included in this study because it is a bilateral task
* Braced and prosthesis wearing groups will greater shoulder abduction and lesser shoulder flexion due to the limitations of the forearm and wrist.
* Shoulder and elbow joint forces and torques will be greater on the sound hand for the amputee group because they will used the prosthesis only as a guide to the task. However, the opposite could occur.

Turning a steering wheel:

* Braced and prosthesis wearing groups will have greater shoulder abduction to compensate for the lack of wrist flexion and extension. However, compensation could also occur in trunk bending.
* For this task the amputee subjects will first complete it with a sound arm and then the prosthesis to determine where compensation occurs.

CONTRIBUTIONS This work will provide many contributions to the biomechanics field and prosthetic design field. One important aspect of studying human maladies is to have a set of control data to use for comparison. Documenting kinematic data of the upper limb during four common tasks will allow for a comparison when studying many upper limb problems or injuries.

This work will help determine if location of new components should be considered in design, fitting and instruction of the upper limb prosthesis. It may also help to bridge the gap between the technological innovation of the engineering field and the clinical astuteness of the prosthetists that are in contact with the end users on a daily basis.

REFERENCES

1. S.C. Jacobsen, D.F. Knutti, R.T. Johnson and H.H. Sears, "Development of the Utah artificial arm," IEEE Trans.Biomed.Eng., vol. 29, pp. 249-269, Apr. 1982.
2. J.E. Uellendahl, "Upper extremity myoelectric prosthetics," Phys.Med.Rehabil.Clin.N.Am., vol. 11, pp. 639-652, Aug. 2000.
3. C.M. Light, P.H. Chappell, B. Hudgins and K. Engelhart, "Intelligent multifunction myoelectric control of hand prostheses," J.Med.Eng.Technol., vol. 26, pp. 139-146, Jul-Aug. 2002.
4. P.J. Kyberd, D.J. Beard and J.D. Morrison, "The population of users of upper limb prostheses attending the Oxford Limb Fitting Service," Prosthet.Orthot.Int., vol. 21, pp. 85-91, Aug. 1997.
5. W. Daly, "Upper extremity socket design options," Phys.Med.Rehabil.Clin.N.Am., vol. 11, pp. 627-638, Aug. 2000.
6. H.H. Sears and J. Shaperman, "Proportional myoelectric hand control: an evaluation," Am.J.Phys.Med.Rehabil., vol. 70, pp. 20-28, Feb. 1991.
7. D.J. Atkins, Heard D. and W.H. Donovan, "Epidemiologic Overview of Individuals with Upper-Limb Loss and Their Reported Research Priorities," JPO, vol. 8, pp. 2-11, 1996. 1996.
8. J.S. Rietman, K. Postema and J.H. Geertzen, "Gait analysis in prosthetics: opinions, ideas and conclusions," Prosthet.Orthot.Int., vol. 26, pp. 50-57, Apr. 2002.
9. M. Twiste and S. Rithalia, "Transverse rotation and longitudinal translation during prosthetic gait--a literature review," J.Rehabil.Res.Dev., vol. 40, pp. 9-18, Jan-Feb. 2003.
10. R.W. Selles, J.B. Bussmand, L.M. Klip, B. Speet, A.J. Van Soest, H.J. Stam, "Adaptations to Mass Perturbations in Transradial Amputees: Kinetic or Kinematic Invariance?," Arch. Phys. Med. Rehabil., vol. 85, pp. 2046-2052, Dec. 2004.
11. A. Murgia, P.J. Kyberd, P.H. Chappell and C.M. Light, "Marker placement to describe the wrist movements during activities of daily living in cyclical tasks," Clin.Biomech.(Bristol, Avon), vol. 19, pp. 248-254, Mar. 2004.
12. R. Safaee-Rad, E. Shwedyk, A.O. Quanbury and J.E. Cooper, "Normal functional range of motion of upper limb joints during performance of three feeding activities," Arch.Phys.Med.Rehabil., vol. 71, pp. 505-509, Jun. 1990.
13. J.S. Landry, "Optimal Fixed Wrist Alignment For Below-Elbow, Powered , Prosthetic Hands," pp. 1-80, 2000. 2000.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-60 years old
* Control group: normal, healthy volunteers
* Amputee group: unilateral, transradial myoelectric prosthesis users

Exclusion Criteria:

* elderly > 60
* children < 18
* pregnant women
* persons with shoulder impairments, injuries, or problems
* bilateral upper limb amputees

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
shoulder abduction
shoulder flexion
elbow flexion
shoulder joint force
should joint torque
elbow joint force
elbow joint torque

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie L Carey, PhD, Principal Investigator — University of South Florida
Locations (1):
- University of South Florida, Tampa, Florida, United States